CLINICAL TRIAL: NCT01591278
Title: Clinical and Radiographic Outcomes of MTA and Biodentine in Pulpotomized Primary Molars. A Randomized Clinical Trial
Brief Title: MTA and Biodentine in Pulpotomized Primary Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cristina Cuadros (Other)
Responsible Party: Sponsor-Investigator, Cristina Cuadros, Cristina Cuadros Fernández, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIC-ODP-1
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Primary Molar Pulpotomy
MeSH Terms: interventions — Pulpotomy; tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulp dressing agent (Experimental)
  Interventions: Other: Pulpotomy
- Pulp dressing (Active Comparator): MTA
  Interventions: Other: Pulpotomy

INTERVENTIONS:
Other: Pulpotomy — Comparison of two different pulp dressing agents
  Arms: Pulp dressing
Other: Pulpotomy — Comparison of two different pulp dressing agents
  Other Names: Biodentine
  Arms: Pulp dressing agent

SUMMARY:
The objective of the study is to evaluate and compare, clinically and radiographically,the effects of MTA and Biodentine when used as pulp dressings following pulpotomy in human primary molars.

ELIGIBILITY:
Inclusion Criteria:

* molars showing:

  1. symptomless exposure of vital pulp by caries
  2. no clinical or radiographic evidence of pulp degeneration (excessive bleeding from the root canal, internal root resorption, inter-radicular and/or furcal bone destruction)
  3. the possibility of proper restoration of the teeth
  4. no physiological resorption of more than one-third of the root

Exclusion Criteria:

* presence of systemic pathology and any history of allergic reaction to latex, local anaesthetics or to the constituents of the test pulp dressing agents

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Number of molars with clinical success | 12 months
Number of molars with radiographic success | 6 and 12 months

SECONDARY OUTCOMES:
Number of molars with no evidence of radicular radiolucency | 6 and 12 months
Number of molars with no evidence of internal resorption | 6 and 12 months
Number of molars with no evidence of external resorption | 6 and 12 months
Number of molars with no evidence of furcation radiolucency | 6 and 12 months
Number of molars with no symptoms of pain | 6 and 12 months
Number of molars without swelling | 6 and 12 months
Number of molars without fistulation | 6 and 12 months
Number of molars without pathological mobility. | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Background] Erdem AP, Guven Y, Balli B, Ilhan B, Sepet E, Ulukapi I, Aktoren O. Success rates of mineral trioxide aggregate, ferric sulfate, and formocresol pulpotomies: a 24-month study. Pediatr Dent. 2011 Mar-Apr;33(2):165-70. PMID 21703067
- [Background] Laurent P, Camps J, About I. Biodentine(TM) induces TGF-beta1 release from human pulp cells and early dental pulp mineralization. Int Endod J. 2012 May;45(5):439-48. doi: 10.1111/j.1365-2591.2011.01995.x. Epub 2011 Dec 22. PMID 22188368
- [Background] Nadin G, Goel BR, Yeung CA, Glenny AM. Pulp treatment for extensive decay in primary teeth. Cochrane Database Syst Rev. 2003;(1):CD003220. doi: 10.1002/14651858.CD003220. PMID 12535462
- [Background] Ansari G, Ranjpour M. Mineral trioxide aggregate and formocresol pulpotomy of primary teeth: a 2-year follow-up. Int Endod J. 2010 May;43(5):413-8. doi: 10.1111/j.1365-2591.2010.01695.x. PMID 20518934
- [Background] Doyle TL, Casas MJ, Kenny DJ, Judd PL. Mineral trioxide aggregate produces superior outcomes in vital primary molar pulpotomy. Pediatr Dent. 2010 Jan-Feb;32(1):41-7. PMID 20298652